CLINICAL TRIAL: NCT04494906
Title: Effects of Interactive Stepping Exercise on Balance and Cognitive Function in Individuals With Parkinson's Disease
Brief Title: Interactive Stepping Exercise on Balance and Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM109104F
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Parkinson's Disease
Keywords: Interactive stepping exercise; Square stepping exercise; Parkinson's disease; Balance ability; Cognitive function
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive stepping exercise group (Experimental): Participants will execute interactive stepping exercise 2 times per week for 8 weeks (16 sessions).
  Interventions: Other: Interactive stepping exercise
- Square stepping exercise group (Active Comparator): Participants will execute square stepping exercise 2 times per week for 8 weeks (16 sessions).
  Interventions: Other: Square stepping exercise

INTERVENTIONS:
Other: Interactive stepping exercise — An exercise intervention based on the principle of square stepping exercise
  Arms: Interactive stepping exercise group
Other: Square stepping exercise — Square stepping exercise
  Arms: Square stepping exercise group

SUMMARY:
The objective of this study is to investigate the effects of interactive stepping exercise on balance and cognitive function in individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD
* Hoehn & Yahr stage between 1 to 3
* Age between 50 to 85
* Stable pharmacologic treatment for the last 2 weeks
* Ability to walk 10 meters unassisted or with assistive devices

Exclusion Criteria:

* Other neurological disorders diagnosis than PD
* Receiving any neurological surgeries
* Any musculoskeletal disorder or cardiopulmonary disease that may influence participation in the study
* The Mini-Mental State Examination (MMSE) < 24 scores
* Participated in other exercise intervention of study in the past 3 months
* Colorblindness or color vision deficiency

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Romberg test | Change from baseline at 8 weeks and 12 weeks
  To evaluate static balance ability
Sharpened Romberg test | Change from baseline at 8 weeks and 12 weeks
  To evaluate static balance ability
One-leg stance test | Change from baseline at 8 weeks and 12 weeks
  To evaluate static balance ability
Timed up and go test | Change from baseline at 8 weeks and 12 weeks
  To evaluate functional walking ability
Mini-Balance Evaluation Systems Test | Change from baseline at 8 weeks and 12 weeks
  To evaluate balance ability
Montreal Cognitive Assessment Chinese version | Change from baseline at 8 weeks and 12 weeks
  To evaluate global cognitive function
Digit span test | Change from baseline at 8 weeks and 12 weeks
  To evaluate executive function
Stroop color and word test Chinese version | Change from baseline at 8 weeks and 12 weeks
  To evaluate executive function
Trail-making test Chinese version | Change from baseline at 8 weeks and 12 weeks
  To evaluate executive function
Spatial span test | Change from baseline at 8 weeks and 12 weeks
  To evaluate visuospatial ability

SECONDARY OUTCOMES:
10-meter walk test | Change from baseline at 8 weeks and 12 weeks
  To evaluate walking ability
Parkinson's Disease Questionnaire 39 | Change from baseline at 8 weeks and 12 weeks
  To evaluate the quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan